CLINICAL TRIAL: NCT01172262
Title: Task-Based Functional MRI (fMRI) Exploration of the Cortical Attention Network in Patients With Severely Bothersome Tinnitus
Brief Title: Task-Based Functional MRI (fMRI) in Patients With Severely Bothersome Tinnitus
Status: Withdrawn | Type: Observational
Why Stopped: Study did not recieve funding, currenlty undergoing protocol revision.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: AMW04292010; Bothersome Tinnitus (Other: Washington University)
Record Dates: First submitted 2010-07-23; First posted 2010-07-29 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Tinnitus
Keywords: Tinnitus; MRI; fMRI; task based MRI; Otolaryngology
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bothered Tinnitus: Either responds with a Global Tinnitus Scale of Moderately or Severely Bothered. Score >30 on the Tinnitus Handicap Index (THI).
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — This is an observational study, no intervention will occur.
  Other Names: This is an observational study, no intervention will occur.

SUMMARY:
Tinnitus is a poorly understood symptom that is often described either as ringing, clicking, ocean sounds, or nature sounds. There is no cure for tinnitus. Approximately 50 million Americans are affected with a small minority being severely affected. This study targets patients with tinnitus who are severely bothered. Through MRI the investigators plan to evaluate the cortical networks of the brain in hopes to better understand this complex process.

DETAILED DESCRIPTION:
Tinnitus is the perceived sensation of sound without actual acoustic stimulation that affects 50 million Americans, with 15 million being significantly bothered. Using functional connectivity MRI (fcMRI), the investigators have found distinct differences in the cortical attention networks between patients with bothersome tinnitus and age-matched controls. These novel findings suggest that some of the classic and most disturbing characteristics of tinnitus result from derangements in cortical pathways. Using a validated task-based functional MRI (fMRI) paradigm developed at Washington University, the investigators will explore the ventral and dorsal frontoparietal cortical attention networks in patients with bothersome tinnitus and non-tinnitus controls.

This will be an experimental task-based fMRI pilot study involving the neurocognitive and neuroimaging assessment of patients with severely bothersome tinnitus.

The investigators plan to perform a pilot study and enroll a total of 10 subjects to undergo task-based imaging. These results will be compared to a control (no tinnitus) cohort (n=35) that has already undergone task-based fMRI. This task-based paradigm will allow us to advance knowledge about the role of the attention, control, and other cortical networks in the development and maintenance of bothersome tinnitus.

The investigators anticipate it will take one year to successfully enroll and test a total of 10 patients. All scans will be performed on the Washington University grounds.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 to 60 years
* Subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater
* Either "moderately bothered" or "severely bothered" on the Global Bothersome scale
* Able to give informed consent
* Able to read, write, speak and understand English fluently
* If applicable, a negative urine pregnancy test
* An audiogram within the past 12 months
* THI score >38

Exclusion Criteria:

* Patients experiencing tinnitus related to cochlear implantation, retrocochlear lesion, Ménière's Disease, or other known anatomic lesions of the ear and temporal bone
* Patients with hyperacusis or misophonia (hyper-sensitivity to noises)
* Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, or any other contraindication for MRI scan
* Patients with an acute or chronic unstable medical condition which, in the opinion of the investigator, would require stabilization prior to initiation of magnetic stimulation
* Patients with any active ear disease that, in the opinion of the PI, needs to be further evaluated
* Patients with symptoms of depression as evidenced by a score of 14 or greater on the Beck Depression Inventory
* Any psychiatric co-morbidity that may complicate the interpretation of study results
* Any tinnitus related to a Workman's Compensation claim or litigation-related event
* Weight over 300 pounds
* A Mini-Mental Status Exam score less than 27
* Patients with a history of claustrophobia
* Inability to lay flat for 2 hour
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year
* Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk
* Unable to provide informed consent
* Currently pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is an observation study focusing on people who have tinnitus and are severely bothered. Recruit a total of 10 participants, preference given to those who live close to 63110.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Perform task based functional imaging on severely bothered tinnitus patients | Analysis will begin after a participant is finished with the study, we anticipate two weeks per patient for complete analysis. Multiple patients can be analyzed at concurrently.
  By undergoing a task based function MRI, we are able to delineate the various attention networks involved with tinnitus. By isolating these networks, insight will be gained on why bothered tinnitus patients have such difficutly.

SECONDARY OUTCOMES:
Perform neurocognitive testing on severely bother tinnitus patients | Analysis will begin after a participant is finished with the study, we anticipate two weeks per patient for complete analysis. Multiple patients can be analyzed at concurrently.
  Through our previously experiences, we have found that those patients with severely bothersome tinnitus have difficulty with neurocognitive testing involving memory and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Wineland, MD, Principal Investigator — Washington University School of Medicine